CLINICAL TRIAL: NCT02286232
Title: A Randomized Trial Comparing a Stretching/Exercise Program and Learning About Self-care Practices From a Self-care Book for Chronic Low Back Pain
Brief Title: Chronic Low Back Pain Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stamford Hospital (Other)
Collaborators: Wilton Family YMCA (Unknown); New Canaan Community YMCA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-0610.01
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic low back pain; stretching exercises
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stretching exercise (Experimental): A series of 12 standardized, weekly stretching exercise classes will be held at the Wilton Family YMCA, designed for people with chronic low back pain unaccustomed to stretching. Participants will be asked to practice the identical routine of that week's stretching exercise class on off days and will be given handouts and CD's to assist in this.
  Interventions: Behavioral: Stretching exercise
- Self-care book (Active Comparator): The Back Pain Helpbook (Moore JE, Lorig K, Von Korff M, Gonzalez VM, Laurent DD. The Back Pain Helpbook. Reading, MA: Perseus Books; 1999)provides information on the causes of back pain and advice on exercising, making appropriate lifestyle modifications, and managing flare-ups.
  Interventions: Behavioral: Self-care book

INTERVENTIONS:
Behavioral: Stretching exercise — This program begins with 10 stretches/exercises over 15 minutes on the initial class and incrementally increases by 1 stretch/exercise each session for a total of 21 stretches/exercises over 30 minutes on the 12th session. The program is designed to stretch/exercise the major muscle groups, emphasizing the neck and arms, trunk, and legs. In addition to the stretches, each class will include breathing exercises and guided imagery for relaxation. Classes will be taught by Physical Therapists who are trained to lead classes through the protocol.
  Arms: Stretching exercise
Behavioral: Self-care book — The Back Pain Helpbook which provides information on the causes of back pain and advice on exercising, making appropriate lifestyle modifications, and managing flare-ups.
  Arms: Self-care book

SUMMARY:
Chronic low back pain is a common condition that can negatively impact quality of life and that lacks highly effective treatment options. The YMCA developed different iterations of a stretching exercise program as a community based treatment for low back pain from 1974-2004. Though anecdotally successful, the YMCA stretching exercise program(s) was not scientifically evaluated for efficacy and became obsolete. The purpose of the study is to test the efficacy of a previously popular YMCA stretching exercise program(s) for back pain. The stretching exercise program that will be studied is a collection of all the resources available for the YMCA stretching exercise program(s). The most recent criteria from a National Institutes of Health sponsored Task Force to study chronic low back pain were applied to this study.

DETAILED DESCRIPTION:
The study will employ a two arm parallel group stratified controlled trial. Statistics were prospectively formulated to compare outcomes of 60 people who completed the study, 30 participants in each intervention group. Subjects from 18 through 64 years old with low back pain on at least half the days over the previous 6 months will be recruited by the Wilton Family YMCA and New Canaan Community YMCA to participate in the study. The participants within each recruitment cohort will be randomized by a sub-investigator who is a statistician to the two treatment arms in a ratio of 1:1 (stretching exercise experimental arm: self-care book active comparator arm). Seven cohorts will receive the intervention stretching exercise program at the Wilton Family YMCA and New Canaan Community YMCA from January 2015 to December 2017. The stretching exercise program consists of 12 standardized weekly stretching exercise sessions that incrementally increase in duration from 15-30 minutes. Participants who receive the stretching exercise intervention will be asked to practice the identical stretches that they did in class on non-class days and will be given handouts and a companion CD to assist in this. Thirty control subjects will receive a self-care book. All analyses will be conducted assuming intent-to-treat principles using SAS statistical software. All P values and 95% CIs will be 2-sided with statistical significance at the P = 0.05 value.

ELIGIBILITY:
Inclusion Criteria:

* Adults from 18 through 64 years old who have had low back pain on at least half the days over the previous 6 months

Exclusion Criteria:

* We will exclude persons whose back pain is attributed to systemic or specific disease such as known cancer, spinal infection, fracture, or ankylosing spondylitis.
* Patients with complex conditions will not participate in the study (eg, sciatica, medicolegal issues, or a previous back surgery).
* We will also exclude persons who do not speak English.
* Finally, persons who are unable to attend classes or unwilling to do home practice will be excluded.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
>=50% improvement in Roland-Morris Disability Questionnaire (RDQ) | 12 weeks after start of study
  RDQ is a widely used health status measure for low back pain. Scale is from 0 (least disability) to 24 (most disability)

SECONDARY OUTCOMES:
>=50% improvement in average pain over previous week from 0-10 scale | 12 weeks after start of study
  0 (no pain) - 10 (worst imaginable pain)
All items derived from PROMIS and STarTBack as suggested by the NIH Task Force | 6, 12, and 24 weeks after start of study
  Composite outcomes of parameters of pain, function, and global assessment as recommended by the NIH Task Force on Research Standards for Low Back Pain
Roland-Morris Disability Questionnaire (RDQ) | 6 and 24 weeks after start of study
  Scale is from 0 (least disability) to 24 (most disability)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Brodsky, MD, Principal Investigator — Stamford Hospital
Locations (1):
- Stamford Hospital, Stamford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No